CLINICAL TRIAL: NCT02458196
Title: A Randomized Trial of Treatment in Patients With IgG4-Related Disease
Brief Title: Study of Treatment Response on IgG4 Related Disease (IgG4RD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgG4-02
Record Dates: First submitted 2015-04-15; First posted 2015-06-01 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-12

CONDITIONS: Autoimmune Disease
Keywords: IgG4 related disease; IgG4-RD; Response rate; Relapse
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease; Recurrence | interventions — Prednisone; prednylidene; Prednisolone; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Prednisone: started with prednisone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, maintained at 7.5mg to 10mg/d to 12 months.
  Interventions: Drug: Prednisone
- Prednisone and Mycophenolate mofetil (Experimental): Prednisone: started with prednisone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, maintained at 7.5mg to 10mg/d to 12 months.
  Immunosuppressive drugs: Mycophenolate mofetil 1g/d-1.5g/d for 6 months and 0.5/d-1.0g/d for 6 months.
  Interventions: Drug: Prednisone and Mycophenolate mofetil

INTERVENTIONS:
Drug: Prednisone — Prednisone: started with prednisone alone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, and maintained at 10mg/d to 12 months.
  Other Names: Pred; Prednisolone
  Arms: Prednisone
Drug: Prednisone and Mycophenolate mofetil — Prednisone: started with prednisone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, maintained at 7.5mg to 10mg/d to 12 months.
  Immunosuppressive drugs: Mycophenolate mofetil 1g/d-1.5g/d for 6 months and 0.5/d-1.0g/d for 6 months.
  Other Names: MMF; Mycophenolate mofetil Dispersible Tablets
  Arms: Prednisone and Mycophenolate mofetil

SUMMARY:
This is an open-label randomized controlled trial to compare the efficacy of Prednisone alone and combination therapy of Prednisone and Mycophenolate mofetil in IgG4RD patients.

DETAILED DESCRIPTION:
Patients with IgG4-RD will be randomized in two therapeutic groups: Prednisone alone and combination therapy with Prednisone and Mycophenolate mofetil. These patients will be followed in 12 months. Treatment response and relapse will be recorded, as well as side effects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18 to 70 years old with informed consent
* All patients must meet the following diagnostic criteria of IgG4RD (2011):

  1. swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sialadenitis (Mikulicz disease), sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions;
  2. elevated serum IgG4 (>1.35 g/L);
  3. histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed). Patients fulfill 1)+2)+3) are diagnosed as definite IgD4RD, 1)+2): possible IgG4RD; 1)+3): probable IgG4RD;
  4. exclusion of other diseases.

Exclusion Criteria:

* Patients will not be included if meets any of the following criteria:

  1. Patients who were diagnosed as other autoimmune diseases;
  2. Patients who were diagnosed as malignant diseases;
  3. Pregnant and lactating women；
  4. Active infection: HIV, HCV, HBV, TB；
  5. Serious organ function failure, expected life time less than 6 months.
  6. Presenting with Mikulicz disease without other manifestations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Complete and partial response rate at 3, 6, 9 and 12 months. | Up to 12 months
  Complete and partial response are defined as resolution of clinical manifestations, biochemical tests (C-reactive Proteins and IgG or IgG4 levels), and imaging studies

SECONDARY OUTCOMES:
Disease response at 3, 6, 9 and 12 months. | Up to 12 months
  Disease response is measured by IgG4-RD Responder Index(IgG4-RD RI) and defined as:
  * Improvement of >2 points in the IgG4-RD RI over baseline
  * No disease flares, as assessed by the IgG4-RD RI.
Number of participants with adverse effect | Up to 12 months
  Treatment-related adverse effect, including glucocorticoid-induced diabetes mellitus and infections.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, Professor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yunyun F, Yu P, Panpan Z, Xia Z, Linyi P, Jiaxin Z, Li Z, Shangzhu Z, Jinjing L, Di W, Yamin L, Xiaowei L, Huadan X, Xuan Z, Xiaofeng Z, Fengchun Z, Yan Z, Wen Z. Efficacy and safety of low dose Mycophenolate mofetil treatment for immunoglobulin G4-related disease: a randomized clinical trial. Rheumatology (Oxford). 2019 Jan 1;58(1):52-60. doi: 10.1093/rheumatology/key227. PMID 30124952